CLINICAL TRIAL: NCT03601936
Title: User Testing Protocol to Evaluate Performance of the Evivo Infant Gut Bifidobacterium Screening Test
Brief Title: User Testing of the Evivo Screening Test
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Additional in-house analysis and development
Sponsor: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EV-8601
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Infants less than 6 months of age (Other): The Evivo Infant Gut Bifidobacterium Screening Test study is a single-group interventional study of 600 female and male infants who are less than 6 months of age and generally healthy.
  Interventions: Device: Evivo Infant Gut Bifidobacterium Screening Test

INTERVENTIONS:
Device: Evivo Infant Gut Bifidobacterium Screening Test — Operators at each test site will collect and test infant stool specimens according to the Evivo Infant Gut Bifidobacterium Screening Test protocol.

SUMMARY:
The study is an evaluation of the Evivo Screening Test's ability to differentiate between high and low levels of Bifidobacterium in infant stool specimens.

DETAILED DESCRIPTION:
This is a prospective, multi-center clinical study of the Evivo Infant Gut Bifidobacterium Screening Test ("Evivo Screening Test").

Lower levels of bifidobacteria in the infant gut have been linked to increased incidence of metabolic and inflammatory disorders. This CLIA Waiver User Testing study is being conducted to evaluate the performance of the Evivo Infant Gut Bifidobacterium Screening Test, which was designed to differentiate between high and low levels of Bifidobacterium in infant stool. This study is intended to confirm the precision of results for this screening test, as well as its ease of use, in a setting that closely resembles the conditions of intended use, specifically the circumstances of sample collection, the location of test sites, and the potential operators.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0-6 months.
* Generally healthy infants.

Exclusion Criteria:

* Infants should not have an acute infection.
* Not intended for use with stool containing meconium.
* Infants with jaundice should not be tested until it has resolved.
* This test should not be used for infants with carbohydrate malabsorption syndrome, which may present with one or more of the following persistent signs: abnormally foul-smelling, mucus-containing, and/or green frothy stools.

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 231 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the Evivo Screening Test's ability to differentiate between high and low levels of Bifidobacterium in infant stool specimens compared to molecular methods (quantitative PCR). | 2 - 6 weeks
  The primary objective of this CLIA Waiver User Testing study is to evaluate the performance of the Evivo Infant Gut Bifidobacterium Screening Test in a setting that closely resembles the conditions of intended use, specifically the circumstances of sample collection, the location of test sites, and the potential operators.

SECONDARY OUTCOMES:
Ease of use of the Evivo Screening Test by operators. | 2 - 6 weeks
  Operators will be asked to complete Operator Questionnaires about their experience using the Screening Test. A 5-point Likert scale will be used to measure outcomes (1 for strongly disagree and 5 for strongly agree). Lower values will represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Flannery, Study Director — rflannery@evolvebiosystems.com
Locations (5):
- United States (5):
  - Matrix Clinical Research, Inc., Los Angeles, California
  - Breastfeed Atlanta LLC, Marietta, Georgia
  - Cyn3rgy Research, Gresham, Oregon
  - Swarthmore Pediatrics, Swarthmore, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided